CLINICAL TRIAL: NCT05254769
Title: Neurofeedback Intervention in Children With Autism Spectrum Disorder (ASD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Collaborators: Khyber Medical University Peshawar (Other)
Responsible Party: Principal Investigator, Dr. Shemaila Saleem, Associate Professor, Shaheed Zulfiqar Ali Bhutto Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFB
Record Dates: First submitted 2022-02-07; First posted 2022-02-24 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Neurofeedback; Autistic Disorder; Autism Spectrum Disorder; Neurodevelopmental Disorders
Keywords: Neurofeedback; Autism Spectrum Disorder
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Neurodevelopmental Disorders

STUDY DESIGN:
Intervention Model Description: Single arm Pre and Post intervention Design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Neurofeedback Intervention in children with Autism Spectrum Disorder (Experimental): Neurofeedback therapy will be provided to 35 children with Autism Spectrum Disorder 30 sessions each and cognitive domains will be assessed before and after intervention.
  Interventions: Device: Neurofeedback Equipment (Cygnet) by BEE Medic GmbH Technologies, Baden-Wurttemberg, Germany.

INTERVENTIONS:
Device: Neurofeedback Equipment (Cygnet) by BEE Medic GmbH Technologies, Baden-Wurttemberg, Germany. — The EEG NeuroAmp (Electroencephalogram Amplifier) is a user-friendly high-performance interface between client and clinician computer. It can be used in two different functionalities: In an EEG/ERP (Event related potential) measurement and in an EEG biofeedback (neurofeedback) and/or peripheral biofeedback setting.

SUMMARY:
This project aims to:

* explore the effectiveness of Neurofeedback therapy for children diagnosed with Autism Spectrum Disorder (ASD)
* assess if cognitive functions are affected before and after Neurofeedback Intervention

DETAILED DESCRIPTION:
Neurofeedback is a computer assisted programmed technique that functions by tracing brain electrical activity (EEG) and providing feedback about the brain activity and sends visual and acoustic signals to counter the mismatch in the electrical activity for improvement. It is a course of learning that allows the patient to observe, regulate and modify his/her own brain activity. Neurofeedback will be carried out in 35 children with Autism Spectrum Disorder (ASD) over a 30-session training period to improve the cognitive functions. This study aims to improve the behavioural and cognitive functions of children and adolescents with Neurofeedback therapy. As Neurofeedback therapy is a non-invasive treatment with almost no side effects, this study will contribute to practice of effective and scalable assessment and treatment strategy for children and adolescents with ASD, utilizing objective tools that have not widely been used in the assessment of Cognitive functions for ASD.

Goal is to improve the quality of life of children on the spectrum by enabling them to perform day to day activities of life and to improve their social communication. Moreover, this study seeks to be a contribution for creating mass awareness regarding the efficacy of Neurofeedback therapy especially in the developing world. Hopefully in the future Neurofeedback training would be incorporated as a standard of care for ASD.

ELIGIBILITY:
Inclusion Criteria:

* 7 to 17 year olds (diagnosed by their physician with autism, in accordance with DSM-V (Diagnostic Statistical Manual-V) diagnostic criteria

Exclusion Criteria: Any child with a history of

* Brain injury
* Bipolar Disorder
* Tourette's Syndrome
* Uncontrolled seizure disorder
* Major psychiatric disorder
* Children on medications

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Childhood Autism Rating Scale (CARS) | Baseline
  Childhood Autism Rating Scale (CARS) is designed as a clinical rating scale for trained clinician to rate items indicative of Autism Spectrum Disorder (ASD) after direct observation of child.The form is used with individuals of all ages and in both clinical and research settings.
IQ (Intelligence Quotient) scoring (Colored Progressive Matrices (CPM) | Baseline
  Tests have been designed to measure as unambiguously as possible, educative and reproductive abilities. It is designed for use with young children and old people, or for those with poor language skills for whatever reason.
Reward sensitivity testing | Baseline
  Neurofeedback is an operant conditioning so the responsiveness and non- responsiveness of the subjects can be attributed to the reward sensitivity. Reward sensitivity for children and adolescents with autism will be assessed by Reward Responsiveness Scale.

SECONDARY OUTCOMES:
Changes in Flanker Inhibitory Control and Attention Score | Baseline, at 10 weeks and 18 weeks
  Flanker Inhibitory Control and Attention Score measures the allocation of one's limited capacities to deal with an abundance of environmental stimulation. It is an assessment of attention and executive Function It will be used to investigate if Neurofeedback therapy affect it and how much. Flanker Inhibitory Control and Attention Score measures the allocation of one's limited capacities to deal with an abundance of environmental stimulation. It is an assessment of attention and executive Function It will be used to investigate if Neurofeedback therapy affect it and to what extent.
Changes in Dimensional Change Card Sort Score; Cognitive Flexibility | Baseline, at 10 weeks and 18 weeks
  Dimensional Change Card Sort Score measures the capacity to plan, organize and monitor the execution of behaviours that are strategically directed in a goal-oriented manner. It is also an assessment of executive functions.
  It will be used to investigate if Neurofeedback therapy affects it and to what extent.
Changes in List Sorting Working Memory Score | Baseline, at 10 weeks and 18 weeks
  List Sorting Working Memory Score measures the ability to store information until the amount of information to be stored exceeds one's capacity to hold that information. It is an assessment of working memory It will be used to investigate if Neurofeedback therapy affects it and to what extent.
Changes in Pattern Comparison Processing Speed Score | Baseline, at 10 weeks and 18 weeks
  Pattern Comparison Processing Speed Score assesses the amount of information that can be processed within a certain unit of time. Items are simple so as to purely measure processing speed.
  It will be used to investigate if Neurofeedback therapy affects it and to what extent.

CONTACTS AND LOCATIONS:
Overall Officials: Shemaila Saleem, Principal Investigator — FM&DC, Shaheed Zulfiqar Ali Bhutto Medical University, Islamabad, Pakistan; Hamid Habib, Principal Investigator — Khyber Medical University, Peshawar, Pakistan
Locations (1):
- Federal Medical and Dental College, Shaheed Zulfiqar Ali Bhutto Medical University, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No